CLINICAL TRIAL: NCT05168267
Title: PTSD Treatment for Incarcerated Men and Women: NIMH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2018-0630: NIMH; R34MH118319 (NIH); A538900 (Other: UW Madison)
Record Dates: First submitted 2021-12-08; First posted 2021-12-23 (Actual); Results first posted 2025-04-08 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-03

CONDITIONS: PTSD
Keywords: Group therapy; Incarcerated Individuals
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Intervention Model Description: Participants are assigned to CPT therapy-intervention group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cognitive Processing Therapy (CPT) group (Experimental): Arm = Cognitive Processing Therapy (CPT) Group = 4 groups of 12 (48 total; 24F/24M) receive CPT to treat PTSD
  Interventions: Behavioral: Cognitive Processing Therapy

INTERVENTIONS:
Behavioral: Cognitive Processing Therapy — CPT: a type of cognitive behavioral therapy recommended for the treatment of PTSD. Delivered over 12 sessions with an emphasis on addressing trauma-related cognitions and challenging trauma-related beliefs. Includes homework assignments. For this study, CPT will be conducted in groups.

SUMMARY:
Study examining the feasibility of and psychological response to group Cognitive Processing Therapy (CPT) in incarcerated men and women with Post-traumatic stress disorder (PTSD). The study will be conducted in male and female incarcerated populations and will include 2 groups of 10 individuals for CPT in both populations (i.e., 40 participants total; 20F/20M). The study will run for up to 2 years. Participants can expect to be participating in study for up to 22 weeks.

DETAILED DESCRIPTION:
Overall Study Objectives:

The primary objectives of this project include:

1. Establish the feasibility of group CPT delivery in male and female incarcerated populations with PTSD;
2. Establish the acceptability of group CPT delivery in male and female incarcerated populations with PTSD;
3. Establish feasibility of assessment collection for primary outcome measures, secondary outcome measures, and potential mediators and moderators during a clinical trial examining group CPT delivery in incarcerated settings.

Prior to beginning any study procedures, informed consent will be obtained orally and in writing. During the informed consent process, eligible participants will be provided with detailed information about the study, including their right to refuse or discontinue participation at any time and the fact that their decision to participate or decline will have no bearing on their standing within the criminal justice system.

Potential participants will be contacted by calling them over the phone system within the prison. When they arrive to the private testing room, they are asked if they would like to learn about the study and potentially participate. If so, participants undergo consent.

Eligible participants will first complete the Clinician-Administered PTSD Scale for DSM-5 (PCL-5) to ascertain current PTSD symptomology and diagnosis. Participants will then be assigned to the CPT groups. The CPT groups will engage in 12, 90-minute treatment sessions (18 hours total). CPT group-members are also asked to complete weekly homework (approximately 12 hours total). A maximum of 6 participants will be included in each CPT session. Participants will be notified via institutional mail when they are starting CPT. Participants will be able to continue any ongoing treatment/interventions they are engaged in within the institution. All participants will be asked what treatment groups they are currently enrolled in during the initial screening to examine the possibility of attentional bias within the CPT group (i.e., more frequent interaction leading to treatment outcomes).

In addition to the treatment groups, CPT group members will also complete a pre-treatment testing session two weeks prior to treatment week 1. After treatment session 5, group members will complete mid-testing assessments. Participants will be called down individually to complete these assessments in a private room with a research assistant after completing the 5th therapy session, but before completing the 8th therapy session. CPT group members will then complete post-treatment testing within one week after completing treatment (group session 12). One month after the treatment is completed, group members will complete the first round of follow-up testing. Three months after the treatment is completed, group members will complete the final round of follow-up testing. Post- and one-month follow up- testing will follow the same procedure as pre- and mid-testing. The three month follow-up session will be identical, with the addition of the PCL-5 interview to re-assess PTSD diagnosis. Group members will be asked to complete 18 sessions in total (pre-, mid-, post-, one-month follow-up testing, three month follow-up testing, 12 treatment groups, and 1 post-intervention focus group).

ELIGIBILITY:
Inclusion Criteria:

* Intelligence quotient (IQ) greater than or equal to 70
* 18 years old or older
* Reading level of 4th grade or higher
* stable medication use (same medication for at least one month)
* able and willing to participate in group therapy
* meet PCL-5 criteria for a current PTSD diagnosis within two months of study enrollment
* no scheduled release date before the end of the treatment group

Exclusion Criteria:

* currently enrolled in trauma focused treatment that is historical or involves processing of trauma itself
* no active symptoms of psychosis that would interfere with the individual's ability to participate in the group
* no active suicidal ideation with intent or plan

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2022-06-06 (Actual); Primary Completion 2024-07-31 (Actual); Study Completion 2024-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael R Koenigs, PhD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- Psychiatric Institute and Clinic, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] James, D.J. and L.E. Glaze, Mental health problems of prison and jail inmates, U.S.D.o. Justice, Editor. 2006: Bureau of Justice Statistics Special Report.
- [Background] Egeressy A, Butler T, Hunter M. 'Traumatisers or traumatised': Trauma experiences and personality characteristics of Australian prisoners. Int J Prison Health. 2009;5(4):212-22. doi: 10.1080/17449200903343209. PMID 25757522
- [Background] Campbell CA, Albert I, Jarrett M, Byrne M, Roberts A, Phillip P, Huddy V, Valmaggia L. Treating Multiple Incident Post-Traumatic Stress Disorder (PTSD) in an Inner City London Prison: The Need for an Evidence Base. Behav Cogn Psychother. 2016 Jan;44(1):112-7. doi: 10.1017/S135246581500003X. Epub 2015 Feb 20. PMID 25697197
- [Background] Resick, P.A., C.M. Monson, and K.M. Chard, Cognitive Processing Therapy for PTSD: A Comprehensive Manual. 2016: Guilford Press.
- [Background] Resick PA, Nishith P, Weaver TL, Astin MC, Feuer CA. A comparison of cognitive-processing therapy with prolonged exposure and a waiting condition for the treatment of chronic posttraumatic stress disorder in female rape victims. J Consult Clin Psychol. 2002 Aug;70(4):867-79. doi: 10.1037//0022-006x.70.4.867. PMID 12182270
- [Background] Morgan RD, Winterowd CL. Interpersonal process-oriented group psychotherapy with offender populations. Int J Offender Ther Comp Criminol. 2002 Aug;46(4):466-82. doi: 10.1177/0306624X02464008. PMID 12150085

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 89 participants were consented, 79 were deemed eligible, 69 started group.
Groups:
- Women's Facility Cognitive Processing Therapy (CPT): Arm = Cognitive Processing Therapy (CPT) Group = Womens Facility: 6 groups of 4-6 (35 total) receive CPT to treat PTSD
  Cognitive Processing Therapy: CPT: a type of cognitive behavioral therapy recommended for the treatment of PTSD. Delivered over 12 sessions with an emphasis on addressing trauma-related cognitions and challenging trauma-related beliefs. Includes worksheet assignments. For this study, CPT will be conducted in groups.
- Men's Facility Cognitive Processing Therapy (CPT): Arm = Cognitive Processing Therapy (CPT) Group = Mens Facility: 6 groups of 4-6 (34 total) receive CPT to treat PTSD
  Cognitive Processing Therapy: CPT: a type of cognitive behavioral therapy recommended for the treatment of PTSD. Delivered over 12 sessions with an emphasis on addressing trauma-related cognitions and challenging trauma-related beliefs. Includes worksheet assignments. For this study, CPT will be conducted in groups.
Period: Overall Study
Arm/Group | Women's Facility Cognitive Processing Therapy (CPT) | Men's Facility Cognitive Processing Therapy (CPT)
Started | 35 | 34
Screened | 55 | 47
Consented to Participate | 46 | 43
Eligible to Participate | 43 | 36
Started Intervention | 34 | 34
Participants Providing Data at 1-week Follow up | 31 | 32
Completed | 31 | 32
Not Completed | 4 | 2
Not completed — Withdrawal by Subject | 2 | 1
Not completed — Withdrawn by Therapist | 1 | 1
Not completed — Left Facility | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Women's Facility Cognitive Processing Therapy (CPT) Group: Arm = Cognitive Processing Therapy (CPT) Group = Women's Facility: 6 groups of 4-6 (35 total) receive CPT to treat PTSD
  Cognitive Processing Therapy: CPT: a type of cognitive behavioral therapy recommended for the treatment of PTSD. Delivered over 12 sessions with an emphasis on addressing trauma-related cognitions and challenging trauma-related beliefs. Includes homework assignments. For this study, CPT will be conducted in groups.
- Total: Total of all reporting groups
Arm/Group | Women's Facility Cognitive Processing Therapy (CPT) Group | Men's Facility Cognitive Processing Therapy (CPT) | Total
Number analyzed (Participants) | 35 | 34 | 69
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.09 (10.78) | 39.6 (11.3) | 38.12 (11.23)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35 | 0 | 35
  Male | 0 | 34 | 34
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 2
  Not Hispanic or Latino | 35 | 32 | 67
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Race was measured by facility (men & women)
  Participants
    Womens Facility: American Indian or Alaska Native | 2 | 0 | 2
    Womens Facility: Asian | 0 | 1 | 1
    Womens Facility: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Womens Facility: Black or African American | 3 | 14 | 17
    Womens Facility: White | 28 | 17 | 45
    Womens Facility: More than one race | 1 | 2 | 3
    Womens Facility: Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 35 | 34 | 69
PCL-5 [Mean (Standard Deviation); unit: units on a scale] — Posttraumatic Stress Disorder Checklist for DSM-5 (PCL-5) PTSD symptom severity is measured by PCL-5 questionnaire (scores from 0, no symptoms, to 80, high severity); primary measure of intervention efficacy
  units on a scale | 50.49 (12.29) | 47.26 (10.31) | 48.90 (11.39)
Beck Anxiety Inventory (BAI) [Mean (Standard Deviation); unit: score on a scale] — Anxiety level measured by score on BAI (between 0 to 63, over 30 = severe anxiety); to characterize our baseline sample of participants
  score on a scale | 22.57 (9.72) | 25.03 (9.32) | 23.72 (9.54)
Beck Depression Inventory 2 (BDI-II) [Mean (Standard Deviation); unit: score on a scale] — Depression level measured by score on BDI-II (between 0 to 63, over 40 = severe depression); to characterize the baseline sample of participants
  score on a scale | 30.14 (11.41) | 29.94 (9.17) | 30.04 (10.29)

OUTCOME MEASURES:

1. Primary Outcome: Number and Percentage of Participants That Attend All Offered Cognitive Processing Therapy Sessions
Description: Intervention feasibility measured primarily by participant retention
Time Frame: up to 6 weeks (by the end of 12th session)
Measure: Count of Participants; unit: Participants
Arm/Group | Women's Facility Cognitive Processing Therapy (CPT) | Men's Facility Cognitive Processing Therapy (CPT)
Number analyzed (Participants) | 35 | 34
Participants | 31 | 32

2. Primary Outcome: Change in Self-reported PTSD Symptoms (PCL-5)
Description: PTSD symptom severity is measured by PCL-5 questionnaire (scores from 0, no symptoms, to 80, high severity); primary measure of intervention efficacy. The negative numbers indicate a decrease in symptom severity of the intervention period.
Time Frame: baseline (one week prior to intervention), post-intervention (up to 13 weeks on study)
Population: Participants with baseline and post-intervention data - the negative numbers indicate a decrease in symptom severity of the intervention period.
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Women's Facility Cognitive Processing Therapy (CPT) | Men's Facility Cognitive Processing Therapy (CPT)
Number analyzed (Participants) | 31 | 32
score on a scale | -19.07 [-58 to -13] | -12.94 [-43 to -12.94]

3. Primary Outcome: Mean Scores on the CSQ-8 (Client Satisfaction Questionnaire)
Description: Client treatment acceptability and satisfaction is measured by mean scores on the CSQ-8; Scores are summed across items once. Items 2, 4, 5, and 8 are reverse scored. Total scores range from 8 to 32, with the higher number indicating greater satisfaction.
Time Frame: Post (1 week post-intervention, up to 13 weeks on study)
Population: Participants lost to follow up
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Women's Facility Cognitive Processing Therapy (CPT) | Men's Facility Cognitive Processing Therapy (CPT)
Number analyzed (Participants) | 29 | 32
units on a scale | 28.48 (3.93) | 25.7 (4.74)

4. Secondary Outcome: Percentage of Individuals That Meet Study Inclusion Criteria
Description: Assesses for participant eligibility as secondary measure of intervention feasibility.
Time Frame: baseline (one week prior to intervention)
Population: Screened participants (one week prior to intervention)
Measure: Count of Participants; unit: Participants
Arm/Group | Women's Facility Cognitive Processing Therapy (CPT) | Men's Facility Cognitive Processing Therapy (CPT)
Number analyzed (Participants) | 55 | 47
Participants | 43 | 36

5. Secondary Outcome: Percentage of Eligible Individuals Enrolled in the Study
Description: Assesses for participant interest as secondary measure of intervention feasibility.
Time Frame: up to start of intervention
Population: Eligible participants
Measure: Count of Participants; unit: Participants
Arm/Group | Women's Facility Cognitive Processing Therapy (CPT) | Men's Facility Cognitive Processing Therapy (CPT)
Number analyzed (Participants) | 43 | 36
Participants | 35 | 34

6. Secondary Outcome: Number of Participants Attending Greater Than or Equal to 75% of Sessions (Attendance)
Description: Assesses for participant compliance: participation during session as secondary measure of intervention feasibility.
Time Frame: By the end of final treatment session (up to 12 weeks)
Measure: Count of Participants; unit: Participants
Arm/Group | Women's Facility Cognitive Processing Therapy (CPT) | Men's Facility Cognitive Processing Therapy (CPT)
Number analyzed (Participants) | 35 | 34
Participants | 31 | 30

7. Secondary Outcome: Percentage of Retained Participants That Completed at Least >80% of Assigned Worksheets
Description: Assesses for participant compliance: extent to which participants complied with treatment skill practice
Time Frame: By the end of final treatment session (up to 12 weeks)
Population: Retained participants (up to 12 weeks on study)
Measure: Count of Participants; unit: Participants
Arm/Group | Women's Facility Cognitive Processing Therapy (CPT) | Men's Facility Cognitive Processing Therapy (CPT)
Number analyzed (Participants) | 31 | 32
Participants | 21 | 22

8. Secondary Outcome: Percentage of Session Elements That Were Rated "Present" (Versus "Absent") by a Clinical Supervisor
Description: Higher percentage indicates better adherence to session elements. Assesses for therapist adherence to CPT guidelines as secondary measure of intervention feasibility. For each 12-session intervention, 2 sessions were audio recorded and rated.
Time Frame: By the end of final treatment session (up to 12 weeks)
Population: CPT session elements
Measure: Number; unit: Percentage of session elements present
Units Other Than Participants: CPT session elements
Arm/Group | Women's Facility Cognitive Processing Therapy (CPT) | Men's Facility Cognitive Processing Therapy (CPT)
Number analyzed (Participants) | 35 | 34
Number analyzed (CPT session elements) | 54 | 60
Percentage of session elements present | 87.72 | 85.96

9. Secondary Outcome: Ratings 1-5 by Clinical Supervisors on Quality of Session Elements Delivered by Therapist
Description: Higher ratings indicate higher-quality session element (scores 1-5; 1="poor", 5="excellent) by the clinical supervisors. Competence ratings will be collected for two audio recorded group sessions out of each 12-session intervention. Assesses for therapist compliance as secondary measure of intervention feasibility.
Time Frame: By the end of final treatment session (up to 12 weeks)
Population: Both unique and non-unique but essential items were analyzed. Unique Items = therapeutic tasks specific to delivery of CPT; Essential Items = therapeutic tasks not specific to CPT but essential to the therapeutic process
Measure: Mean (Standard Deviation); unit: CPT session elements
Units Other Than Participants: CPT session elements
Arm/Group | Women's Facility Cognitive Processing Therapy (CPT) | Men's Facility Cognitive Processing Therapy (CPT)
Number analyzed (Participants) | 35 | 34
Number analyzed (CPT session elements) | 54 | 60
CPT session elements
  Unique Items | 4.67 (.57) | 4.35 (.5)
  Essential Items | 4.77 (.43) | 4.36 (.53)

10. Secondary Outcome: Number of Participants Reporting Increased Suicidality Over the Course of Treatment (Endorsing 2 or Higher on Question #9 of BDI-II)
Description: Question 9 on the BDI-II assesses for suicidal ideation. A score of 2 (I would like to kill myself) or 3 (I would kill myself if I had the chance; the highest score) indicate heightened levels of suicidal ideation. Participants who endorse current suicidal ideation will be referred to mental health services within the institution. Assesses for participant safety as secondary measure of intervention feasibility.
Time Frame: post (one week post-intervention, up to 13 weeks on study)
Measure: Count of Participants; unit: Participants
Arm/Group | Women's Facility Cognitive Processing Therapy (CPT) | Men's Facility Cognitive Processing Therapy (CPT)
Number analyzed (Participants) | 35 | 34
Participants | 0 | 2

11. Secondary Outcome: Reasons for Participant Discontinuation
Description: We will collect information on participant dropout reasons to understand reasons for discontinuation
Time Frame: Up to 3 month follow up (up to 25 weeks)
Measure: Count of Participants; unit: Participants
Arm/Group | Women's Facility Cognitive Processing Therapy (CPT) | Men's Facility Cognitive Processing Therapy (CPT)
Number analyzed (Participants) | 35 | 34
Participants
  Transferred Facilities | 1 | 0
  Scheduling Issues | 1 | 0
  Group "Not Helpful" | 1 | 0
  Work | 0 | 2
  Withdrawn by study clinician | 0 | 2

ADVERSE EVENTS:
Time Frame: Adverse events were collected from consented (one week prior to intervention) to the three month follow up (12 weeks after intervention, up to 25 weeks total)
Description: Since this is a mental health study, our definition of an adverse event slightly differs from ClinicalTrials.gov definitions. If the participant exhibits any negative/significant psychological symptoms, social issues, physical injuries, medical injuries, or other negative life events, this is considered an adverse event.
Arm/Group | Women's Facility Cognitive Processing Therapy (CPT) | Men's Facility Cognitive Processing Therapy (CPT)
All-Cause Mortality (participants affected / at risk) | 0/35 | 0/34
Serious Adverse Events (participants affected / at risk) | 0/35 | 0/34
Other Adverse Events (participants affected / at risk) | 7/35 | 14/34
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Women's Facility Cognitive Processing Therapy (CPT) (N=35) | Men's Facility Cognitive Processing Therapy (CPT) (N=34)
Passive Suicidal Ideation (Psychiatric disorders) | 0 (0) | 2 (2)
Increased PTSD symptoms (Psychiatric disorders) | 1 (1) | 3 (3) — Nightmares, Increase in PTSD symptom on PCL-5
Increase in depressive symptoms (Psychiatric disorders) | 0 (0) | 3 (3)
Segregated Housing Placement / Rule Violation (Social circumstances) | 3 (3) | 3 (3)
Medical Event (Cardiac disorders) | 1 (1) | 5 (6) — Hip issue requiring crutches, carpal tunnel syndrome, nerve pain in neck, dizziness and fainting due to existing condition, bedrest for unknown illness, infected finger
Increased emotional distress (Psychiatric disorders) | 2 (2) | 0 (0)
Social Circusmtances (Social circumstances) | 0 (0) | 4 (4) — Family member assaulted, argument with peer, kicked out of school, legal issues

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2025-01-22): https://cdn.clinicaltrials.gov/large-docs/67/NCT05168267/Prot_SAP_ICF_000.pdf